CLINICAL TRIAL: NCT05996497
Title: Evaluation of Speech Rhythm Training in Dyslexic Readers Aged 7 to 9 Years
Acronym: RnDys
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Institut de l'Audition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2022-063; 2022-A01132-41 (Other: ID RCB)
Record Dates: First submitted 2023-05-22; First posted 2023-08-18 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Dyslexia
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Auditory Rhythmic at 30 Hz then GraphoGame (Other): Training 1 with Auditory Rhythmic at 30 Hz (6 weeks) then Training 2 with GraphoGame (6 weeks)
  Interventions: Behavioral: behavioral measures; Other: Electrophysiological measures; Other: Training 1; Other: Training 2
- GraphoGame then Rhythmic Auditory at 30 Hz (Other): Training 1 with GraphoGame (6 weeks) then Training 2 with Auditory Rhythmic at 30 Hz (6 weeks)
  Interventions: Behavioral: behavioral measures; Other: Electrophysiological measures; Other: Training 1; Other: Training 2
- Auditory Rhythmic at low frequencies then GraphoGame (Other): Training 1 with Auditory Rhythmic at low frequencies (6 weeks) then Training 2 with GraphoGame (6 weeks)
  Interventions: Behavioral: behavioral measures; Other: Electrophysiological measures; Other: Training 1; Other: Training 2
- GraphoGame then Auditory Low Frequency Rhythmic (Other): Training 1 with GraphoGame (6 weeks) then Training 2 with Auditory Rhythmic at Low Frequency Rhythmic (6 weeks)
  Interventions: Behavioral: behavioral measures; Other: Electrophysiological measures; Other: Training 1; Other: Training 2

INTERVENTIONS:
Behavioral: behavioral measures — behavioral measures
Other: Electrophysiological measures — Electrophysiological measures
Other: Training 1 — Training 1
Other: Training 2 — Training 2

SUMMARY:
Studies of dyslexia have shown altered oscillatory activity in the low gamma band (~25-35 Hz) in the left auditory cortex. Neural oscillations around 30 Hz constitute the basic sampling rate of speech, from which the ability to form specific phonemic categories on which reading learning is based is derived. An alteration of the oscillatory activity at 30 Hz could therefore influence the ability of children to learn to read, and explain the reading deficit observed in children with a specific written language disorder. The objective of our study is to determine whether intensive rhythmic auditory stimulation applied during 30 sessions of 15 minutes spread over 6 weeks (5 sessions per week) can correct neural oscillations in the gamma-low band, allowing an improvement of phonemic categorization abilities, and thus the reading abilities of dyslexic readers aged 7 to 9 years. The long-term objective of this study is to test the therapeutic potential of auditory stimulation with speech rhythms for the treatment of reading disorders.

DETAILED DESCRIPTION:
Longitudinal cross-over study carried out on 4 experimental groups to compare the effect of two rhythmic auditory trainings (30 Hz and low frequencies) compared to the effect of a grapho-phonological correspondence training (GraphoGame).

The study begins with a recruitment and inclusion period after diagnosis of dyslexia. During this study, 4 assessments are performed and include behavioral measures in the care setting and electrophysiological measures in the research setting:

* at time T1 before any remediation,
* at T2 after the first training,
* at T3 at most 7 days after the 2nd training session,
* at T4 seven weeks after T3.

After the T1 assessment, participants were randomized into 4 different groups (training 1 then training 2):

Group 1 : Auditory Rhythmic at 30 Hz then GraphoGame Group 2 : GraphoGame then Rhythmic Auditory at 30 Hz Group 3 : Auditory Rhythmic at low frequencies then GraphoGame Group 4 : GraphoGame then Auditory Low Frequency Rhythmic The first training period (total duration 6 weeks) according to the assigned group begins and takes place at the speech therapist's office and at home.

After the T2 evaluation, the 2nd training period (total duration 6 weeks) according to the assigned group begins and takes place at the SLP's office as well as at home.

The post-training evaluations T3 and T4 take place, respectively, 1 week and 7 weeks after the last training.

ELIGIBILITY:
Inclusion Criteria:

* between 7 and 9 years old
* in regular schooling
* have a diagnosis of dyslexia
* have a non-verbal intelligence assessment within the norm. Inclusion assessments must show a major reading disability without associated cognitive deficits.
* be equipped with a PC at home
* have given their assent and whose parents/legal guardians have given their oral consent

Exclusion Criteria:

* have any other diagnosis of language impairment
* have a neurological disorder (visual, auditory, executive)
* have an associated psychiatric disorder
* have a developmental delay.

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of reading accuracy by measuring the percentage of correct responses in the isolated pseudoword reading task between rythmic auditory training condition vs. grapho-phonological mapping training (GraphoGame). | 2 years
  Comparison of reading performance is assessed in terms of both accuracy and speed. High percentage of correct responses means that children improve their reading accuracy.
Comparison of reading speed by measuring reading time in the isolated pseudoword reading task between rythmic auditory training condition vs. grapho-phonological mapping training (GraphoGame). | 2 years
  Comparison of reading performance is assessed in terms of both accuracy and speed. A short time means that children improve their reading speed.

SECONDARY OUTCOMES:
Measurement of reading accuracy (percentage of correct responses in the isolated pseudoword reading task) between multiple conditions. | 2 years
  Reading accuracy compared between rhythmic auditory training then grapho-phonological mapping training vs. grapho-phonological mapping training then rhythmic auditory training and rhythmic auditory training at 30 Hz vs. rhythmic auditory training at 3.5 Hz
Measurement of reading speed (reading time in the isolated pseudoword reading task) between multiple conditions. | 2 years
  Reading speed compared between rhythmic auditory training then grapho-phonological mapping training vs. grapho-phonological mapping training then rhythmic auditory training and rhythmic auditory training at 30 Hz vs. rhythmic auditory training at 3.5 Hz

CONTACTS AND LOCATIONS:
Overall Officials: Diane Lazard, MD, Principal Investigator — Institut Pasteur; Anne-Lise Giraud, PhD, Study Director — Institut Pasteur
Locations (1):
- Institut de l'Audition, Paris, France